CLINICAL TRIAL: NCT06529926
Title: Investigation of The Effect of "Instrument-Assisted Soft Tissue Mobilization" in Individuals With Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Muhammed Usame TAS, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ÜSAME TAŞ-004
Record Dates: First submitted 2024-07-21; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Instrument-assisted Soft Tissue Mobilization; Treatment; Exercise; Pain
MeSH Terms: conditions — Motor Activity; Pain | interventions — Watchful Waiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Treated with classical physiotherapy (Hotpack+TENS+Ultrasound) program. A 20-minute hotpack was applied to the lumbar area. TENS and ultrasound were applied as electrotherapy agents. The TENS application was made with the Chattanooga Intelect Advanced Combo device. Conventional tens was applied at a frequency of 100 Hz for 20 min with a current of 100 μs. The ultrasound application was made with the Chattanooga Intelect Advanced Combo device. Lumbar area was administered at a dose of 1 MHz, 1.5 W/cm² using a 5 cm diameter cap for 6 min. In the first session, the physiotherapist had the patient explain the exercises (posterior pelvic tilt exercise, hip flexors stretching exercise, lumbar extensors stretching exercise, abdominal muscle strengthening exercise, SLR exercise, pelvic elevation exercise, cat-camel exercise and lumbar extensor strengthening exercise). Afterwards, patients were advised to rest for 1 minute between exercises, 1 time a day and for 4 weeks, 5 days a week.
  Interventions: Other: Observational
- IASTM Treatment Group (Experimental): IASTM application was applied at an angle of 45° in a direction parallel to the muscle fibers for about 20 seconds. Immediately afterwards, a total of 40 seconds of treatment time was applied by treating the muscle fibers at a 45° angle with the instrument for an additional 20 seconds in a direction perpendicular to them. In other words, for each area (paraspinal muscles, gluteus maximus and gluteus medius muscles, hamstrings), a total of 2 minutes was applied to the right and left sides separately for 40x3 seconds. Paraspinal muscles were treated from caudal to cranium, gluteal muscles from proximal to distal and hamstring muscles from popliteal fossa to gluteal line. Stretching was provided by exercises applied to the control group. After the cold application, IASTM application was made, the cold-pack was applied to each area for 5 minutes. (The application was performed by a trained and experienced physiotherapist and with a stainless steel gua sha device).
  Interventions: Other: IASTM Technique Application

INTERVENTIONS:
Other: Observational — Only classical physiotherapy application for 4 weeks.
  Arms: Control Group
Other: IASTM Technique Application — IASTM application for 2 sessions per week with classical physiotherapy for 4 weeks.
  Arms: IASTM Treatment Group

SUMMARY:
Instrument-assisted soft tissue mobilization is an instrument-assisted soft tissue mobilization technique. It consists of stainless steel instrument designed to adapt to various tissues/shapes/curves of the body. The instruments were developed as an alternative to transverse friction massage. Stainless steel acts a bit like a diaposon when it comes into contact with fibrotic tissue. A resonance or reverberation in the instrument is created upon contact and transmitted through the instrument to the hands of the clinician. The application of heavy pressure (compared to light or medium pressure) using instruments has been proven to promote a greater fibroblastic response.

Instrument-assisted soft tissue mobilization is not used without insulation. It is imperative to use movement and strengthening in combination with soft tissue mobilization to promote tissue adaptation and remodeling. Mechanical loading has been shown to affect chondrocyte alignment and fibroblast activity with increased proteoglycan and collagen synthesis. The aim of this study was to investigate the effects of the IASTM technique on individuals of different ages diagnosed with LDH.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals have been diagnosed with LDH,
2. Their pain is 3 and above according to the Visual Analog Scale (VAS),
3. They are between the ages of 20-60,
4. Their clinical status is stable,
5. They are fully cooperative,
6. They do not have cognitive, cognitive and mental problems and they can express themselves,
7. They voluntarily agree to participate in the study.

Exclusion Criteria:

1. Individuals have psychological disorders, mental disorders, cancer and severe depression,
2. Primary or metastatic spinal malignancy,
3. Have been diagnosed with advanced osteoporosis,
4. Have recently undergone surgical intervention or acute infection,
5. Cannot or do not want to perform tests or treatment exercises,
6. Want to leave voluntarily.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of Pain | Pre-treatment assessment.
  Visual analog scale was used to evaluate the pain of the patients.
Evaluation of Pain | After 4 weeks of treatment (Post-treatment assessment).
  Visual analog scale was used to evaluate the pain of the patients.
Evaluation of Pain | 2nd month post-treatment assessment.
  Visual analog scale was used to evaluate the pain of the patients.
Evaluation of Functional Status (Straight leg raise test) | Pre-treatment assessment.
  Straight leg raise test was used to evaluate the functional status of the patients.
Evaluation of Functional Status (Straight leg raise test) | After 4 weeks of treatment (Post-treatment assessment).
  Straight leg raise test was used to evaluate the functional status of the patients.
Evaluation of Functional Status (Straight leg raise test) | 2nd month post-treatment assessment.
  Straight leg raise test was used to evaluate the functional status of the patients.
Evaluation of Functional Status (Slump test) | Pre-treatment assessment.
  Slump test was used to evaluate the functional status of the patients.
Evaluation of Functional Status (Slump test) | After 4 weeks of treatment (Post-treatment assessment).
  Slump test was used to evaluate the functional status of the patients.
Evaluation of Functional Status (Slump test) | 2nd month post-treatment assessment.
  Slump test was used to evaluate the functional status of the patients.
Evaluation of Functional Status (5-min walking test) | Pre-treatment assessment.
  5-min walking test was used to evaluate the functional status of the patients.
Evaluation of Functional Status (5-min walking test) | After 4 weeks of treatment (Post-treatment assessment).
  5-min walking test was used to evaluate the functional status of the patients.
Evaluation of Functional Status (5-min walking test) | 2nd month post-treatment assessment.
  5-min walking test was used to evaluate the functional status of the patients.
Evaluation of Normal Joint ROM | Pre-treatment assessment.
  Goniometer was used to evaluate the normal joint ROM of the patients.
Evaluation of Normal Joint ROM | After 4 weeks of treatment (Post-treatment assessment).
  Goniometer was used to evaluate the normal joint ROM of the patients.
Evaluation of Normal Joint ROM | 2nd month post-treatment assessment.
  Goniometer was used to evaluate the normal joint ROM of the patients.
Evaluation of Quality of Life | Pre-treatment assessment.
  Short Form-36 was used to evaluate the quality of life of the patients.
Evaluation of Quality of Life | After 4 weeks of treatment (Post-treatment assessment).
  Short Form-36 was used to evaluate the quality of life of the patients.
Evaluation of Quality of Life | 2nd month post-treatment assessment.
  Short Form-36 was used to evaluate the quality of life of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Üsame TAŞ, Lecturer, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No